CLINICAL TRIAL: NCT03704857
Title: Evaluation of the Effectiveness of Different Endodontic Treatment Techniques in Postoperative Symptoms, Apical Repair, Longevity of Rehabilitations, and Oral Health-related Quality of Life
Brief Title: Different Endodontic Treatment Techniques in Postoperative Symptoms, Apical Repair, Longevity of Rehabilitations, and Oral Health-related Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Livia Azeredo Alves Antunes, Clinical professor, Universidade Federal Fluminense
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: Endodontic therapy and symptom
Record Dates: First submitted 2018-08-16; First posted 2018-10-15 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Endodontically Treated Teeth; Postoperative Pain; Edema; Photochemotherapy
Keywords: Root canal Preparation; Foraminal enlargement; Photobiomodulation therapies; Postoperative symptoms; Passive ultrassonic irrigation; Irrigating solutions; Filling materials; Mouth Rehabilitation; Apical repair; Oral health-related quality of life; Antimicrobial photodynamic therapy; Low-level laser therapy
MeSH Terms: conditions — Tooth, Nonvital; Pain, Postoperative; Edema | interventions — Low-Level Light Therapy; Cryotherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Foraminal enlargement with sodium hypochlorite as irrigant (Active Comparator): Unirradicular teeth will be submitted to endodontic treatment with foraminal enlargement, instrumentation with reciprocating rotation, sodium hypochlorite as irrigant, lateral condensation filling with MTA Fillapex. The analysis of the postoperative symptoms will be performed by the visual analog pain scale at 1th, 2th, 3th, 4th, 5th, 6th, 7th, 14th and 30th days and by the clinical evaluation of edema in 48 and 72 hours. The periapical lesion repair will be evaluated clinically and radiographically at 3, 6, 12, 18 and 24 months. The longevity of rehabilitations will be performed clinically and radiographically for 24 months. In addition, patients will respond a quality of life questionnaire (OHIP-14) on the day of endodontic treatment, on the 7th day and on the 30th day.
  Interventions: Other: Foraminal Enlargement / Irrigating solutions / Filling materials; Other: OHIP-14; Other: Assessment of pain and edema; Other: Assessment of periapical lesion; Other: Longevity of rehabilitations
- Foraminal enlargement with sodium hypochlorite and photobiomodulation (Experimental): Unirradicular teeth will be submitted to endodontic treatment with foraminal enlargement, instrumentation with reciprocating rotation, sodium hypochlorite as irrigant, photobiomodulation (antimicrobial photodynamic therapy and low-level laser therapy), lateral condensation filling with MTA Fillapex. The analysis of the postoperative symptoms will be performed by the visual analog pain scale at 1th, 2th, 3th, 4th, 5th, 6th, 7th, 14th and 30th days and by the clinical evaluation of edema in 48 and 72 hours. The periapical lesion repair will be evaluated clinically and radiographically at 3, 6, 12, 18 and 24 months. The longevity of rehabilitations will be performed clinically and radiographically for 24 months. In addition, patients will respond a quality of life questionnaire (OHIP-14) on the day of endodontic treatment, on the 7th day and on the 30th day.
  Interventions: Other: Foraminal Enlargement / Irrigating solutions / Filling materials; Other: Photobiomodulation; Other: OHIP-14; Other: Assessment of pain and edema; Other: Assessment of periapical lesion; Other: Longevity of rehabilitations
- Foraminal enlargement with chlorhexidine as irrigant (Experimental): Unirradicular teeth will be submitted to endodontic treatment with foraminal enlargement, instrumentation with reciprocating rotation, chlorhexidine as irrigant, lateral condensation filling with MTA Fillapex. The analysis of the postoperative symptoms will be performed by the visual analog pain scale at 1th, 2th, 3th, 4th, 5th, 6th, 7th, 14th and 30th days and by the clinical evaluation of edema in 48 and 72 hours. The periapical lesion repair will be evaluated clinically and radiographically at 3, 6, 12, 18 and 24 months. The longevity of rehabilitations will be performed clinically and radiographically for 24 months. In addition, patients will respond a quality of life questionnaire (OHIP-14) on the day of endodontic treatment, on the 7th day and on the 30th day.
  Interventions: Other: Foraminal Enlargement / Irrigating solutions / Filling materials; Other: OHIP-14; Other: Assessment of pain and edema; Other: Assessment of periapical lesion; Other: Longevity of rehabilitations
- Foraminal enlargement with sodium hypochlorite and AH Plus (Active Comparator): Unirradicular teeth will be submitted to endodontic treatment with foraminal enlargement, instrumentation with reciprocating rotation, sodium hypochlorite as irrigant, lateral condensation filling with AH Plus.The analysis of the postoperative symptoms will be performed by the visual analog pain scale at 1th, 2th, 3th, 4th, 5th, 6th, 7th, 14th and 30th days and by the clinical evaluation of edema in 48 and 72 hours. The periapical lesion repair will be evaluated clinically and radiographically at 3, 6, 12, 18 and 24 months. The longevity of rehabilitations will be performed clinically and radiographically for 24 months. In addition, patients will respond a quality of life questionnaire (OHIP-14) on the day of endodontic treatment, on the 7th day and on the 30th day.
  Interventions: Other: Foraminal Enlargement / Irrigating solutions / Filling materials; Other: OHIP-14; Other: Assessment of pain and edema; Other: Assessment of periapical lesion; Other: Longevity of rehabilitations
- Foraminal enlargement with conventional irrigation (Active Comparator): Molars will be submitted to endodontic treatment with foraminal enlargement, instrumentation with reciprocating rotation, conventional irrigation with sodium hypochlorite, lateral condensation filling with MTA Fillapex. The analysis of the postoperative symptoms will be performed by the visual analog pain scale at 1th, 2th, 3th, 4th, 5th, 6th, 7th, 14th and 30th days and by the clinical evaluation of edema in 48 and 72 hours. The periapical lesion repair will be evaluated clinically and radiographically at 3, 6, 12, 18 and 24 months. The longevity of rehabilitations will be performed clinically and radiographically for 24 months. In addition, patients will respond a quality of life questionnaire (OHIP-14) on the day of endodontic treatment, on the 7th day and on the 30th day.
  Interventions: Other: Foraminal Enlargement / Irrigating solutions / Filling materials; Other: OHIP-14; Other: Assessment of pain and edema; Other: Assessment of periapical lesion; Other: Longevity of rehabilitations
- Foraminal enlargement with passive ultrasonic irrigation (Experimental): Molars will be submitted to endodontic treatment with foraminal enlargement, instrumentation with reciprocating rotation, passive ultrasonic irrigation with sodium hypochlorite, lateral condensation filling with MTA Fillapex. The analysis of the postoperative symptoms will be performed by the visual analog pain scale at 1th, 2th, 3th, 4th, 5th, 6th, 7th, 14th and 30th days and by the clinical evaluation of edema in 48 and 72 hours. The periapical lesion repair will be evaluated clinically and radiographically at 3, 6, 12, 18 and 24 months.The longevity of rehabilitations will be performed clinically and radiographically for 24 months. In addition, patients will respond a quality of life questionnaire (OHIP-14) on the day of endodontic treatment, on the 7th day and on the 30th day.
  Interventions: Other: Foraminal Enlargement / Irrigating solutions / Filling materials; Other: Passive ultrasonic irrigation; Other: OHIP-14; Other: Assessment of pain and edema; Other: Assessment of periapical lesion; Other: Longevity of rehabilitations
- Foraminal enlargement with cryotherapy (Experimental): Unirradicular teeth will be submitted to endodontic treatment with foraminal enlargement, instrumentation with reciprocating rotation, sodium hypochlorite as irrigant, cryotherapy with saline solution, lateral condensation filling with MTA Fillapex. The analysis of the postoperative symptoms will be performed by the visual analog pain scale at 1th, 2th, 3th, 4th, 5th, 6th, 7th, 14th and 30th days and by the clinical evaluation of edema in 48 and 72 hours. The periapical lesion repair will be evaluated clinically and radiographically at 3, 6, 12, 18 and 24 months. The longevity of rehabilitations will be performed clinically and radiographically for 24 months. In addition, patients will respond a quality of life questionnaire (OHIP-14) on the day of endodontic treatment, on the 7th day and on the 30th day.
  Interventions: Other: Foraminal Enlargement / Irrigating solutions / Filling materials; Other: OHIP-14; Other: Assessment of pain and edema; Other: Assessment of periapical lesion; Other: Longevity of rehabilitations; Other: Cryotherapy
- Foraminal enlargement with cryotherapy and AH Plus (Experimental): Unirradicular teeth will be submitted to endodontic treatment with foraminal enlargement, instrumentation with reciprocating rotation, sodium hypochlorite as irrigant, cryotherapy with saline solution, lateral condensation filling with AH Plus. The analysis of the postoperative symptoms will be performed by the visual analog pain scale at 1th, 2th, 3th, 4th, 5th, 6th, 7th, 14th and 30th days and by the clinical evaluation of edema in 48 and 72 hours. The periapical lesion repair will be evaluated clinically and radiographically at 3, 6, 12, 18 and 24 months. The longevity of rehabilitations will be performed clinically and radiographically for 24 months. In addition, patients will respond a quality of life questionnaire (OHIP-14) on the day of endodontic treatment, on the 7th day and on the 30th day.
  Interventions: Other: Foraminal Enlargement / Irrigating solutions / Filling materials; Other: OHIP-14; Other: Assessment of pain and edema; Other: Assessment of periapical lesion; Other: Longevity of rehabilitations; Other: Cryotherapy
- Foraminal enlargement with ozone therapy (Experimental): Unirradicular teeth will be submitted to endodontic treatment with foraminal enlargement, instrumentation with reciprocating rotation, sodium hypochlorite as irrigant, ozone therapy, lateral condensation filling with MTA Fillapex. The analysis of the postoperative symptoms will be performed by the visual analog pain scale at 1th, 2th, 3th, 4th, 5th, 6th, 7th, 14th and 30th days and by the clinical evaluation of edema in 48 and 72 hours. The periapical lesion repair will be evaluated clinically and radiographically at 3, 6, 12, 18 and 24 months. The longevity of rehabilitations will be performed clinically and radiographically for 24 months. In addition, patients will respond a quality of life questionnaire (OHIP-14) on the day of endodontic treatment, on the 7th day and on the 30th day.
  Interventions: Other: Foraminal Enlargement / Irrigating solutions / Filling materials; Other: OHIP-14; Other: Assessment of pain and edema; Other: Assessment of periapical lesion; Other: Longevity of rehabilitations; Other: Ozone therapy
- Foraminal enlargement with ozone therapy and AH Plus (Experimental): Unirradicular teeth will be submitted to endodontic treatment with foraminal enlargement, instrumentation with reciprocating rotation, sodium hypochlorite as irrigant, ozone therapy, lateral condensation filling with AH Plus. The analysis of the postoperative symptoms will be performed by the visual analog pain scale at 1th, 2th, 3th, 4th, 5th, 6th, 7th, 14th and 30th days and by the clinical evaluation of edema in 48 and 72 hours. The periapical lesion repair will be evaluated clinically and radiographically at 3, 6, 12, 18 and 24 months. The longevity of rehabilitations will be performed clinically and radiographically for 24 months. In addition, patients will respond a quality of life questionnaire (OHIP-14) on the day of endodontic treatment, on the 7th day and on the 30th day.
  Interventions: Other: Foraminal Enlargement / Irrigating solutions / Filling materials; Other: OHIP-14; Other: Assessment of pain and edema; Other: Assessment of periapical lesion; Other: Longevity of rehabilitations; Other: Ozone therapy

INTERVENTIONS:
Other: Foraminal Enlargement / Irrigating solutions / Filling materials — Instrumentation with foraminal enlargement and various irrigation solutions and filling materials will be performed according to the allocated group.
  The foraminal enlargement provides better results in the bacterial removal of the apical portion of the root canal. This instrumentation will be done with the Reciproc 40 or 50 system in the apical foramen, determined by the apical locator.
  To contribute to disinfection of the root canal, sodium hypochlorite and chlorhexidine are the most widely used irrigators. Sodium hypochlorite has a broad antimicrobial spectrum and an effective ability to dissolve organic matter and necrotic tissue; while chlorhexidine shows substantivity and antimicrobial residual activity when used as an irrigating substance.
  Besides that, MTA Fillapex or AH Plus will be used and the recommended filling technique will be lateral condensation.
Other: Photobiomodulation — aPDT will be performed with 0.01% methylene blue solution and it will be inserted into the root canal for 5 minutes. The excess will be removed and irradiation will be performed inside the root canal with the red laser of Índio Gálio Alumínio Fósforo (660nm, Laser Duo, MMOptics, São Paulo, SP, Brazil) for 90 seconds. Laser therapy with Gallium-Aluminum-Arsenic infrared laser (808nm, Laser Duo, MMOptics, São Paulo, SP, Brazil) will be performed on the gingiva from the vestibular face and on the palatal / lingual face, both located in the periapical region for 40 seconds.
  Arms: Foraminal enlargement with sodium hypochlorite and photobiomodulation
Other: Passive ultrasonic irrigation — PUI will be performed with Newtron P5 ultrasound (Satelec / Acteon Group, Bordeaux, France), at intensity 9 and with a 25mm (# 0.25, taper 0.00). The protocol of use will be 3 sequences of 20 seconds of ultrasonic activation with 2 ml of sodium hypochlorite 2.5% in each root canal.
  Arms: Foraminal enlargement with passive ultrasonic irrigation
Other: OHIP-14 — Patients will respond a quality of life questionnaire (OHIP-14) on the day of endodontic treatment, on the 7th day and on the 30th day.
Other: Assessment of pain and edema — The analysis of the postoperative symptoms will be performed by the visual analog pain scale at 1th, 2th, 3th, 4th, 5th, 6th, 7th, 14th and 30th days and by the clinical evaluation of edema in 48 and 72 hours.
Other: Assessment of periapical lesion — The periapical lesion repair will be evaluated clinically and radiographically at 3, 6, 12, 18 and 24 months.
Other: Longevity of rehabilitations — The teeth will be rehabilitated with resin and glass fiber post. The longevity of rehabilitations will be performed clinically and radiographically for 24 months.
Other: Cryotherapy — The analysis of the postoperative symptoms will be performed by the visual analog pain scale at 1th, 2th, 3th, 4th, 5th, 6th, 7th, 14th and 30th days and by the clinical evaluation of edema in 48 and 72 hours.
  Arms: Foraminal enlargement with cryotherapy; Foraminal enlargement with cryotherapy and AH Plus
Other: Ozone therapy — The analysis of the postoperative symptoms will be performed by the visual analog pain scale at 1th, 2th, 3th, 4th, 5th, 6th, 7th, 14th and 30th days and by the clinical evaluation of edema in 48 and 72 hours.
  Arms: Foraminal enlargement with ozone therapy; Foraminal enlargement with ozone therapy and AH Plus

SUMMARY:
Objective: The objective of this study will be to evaluate the effectiveness of different endodontic treatment techniques in postoperative symptoms, apical repair, longevity of rehabilitations, and oral health-related quality of life.

Methods: This prospective, randomized, double-blind clinical study was approved at the Research Ethics Committee (nº 2.353.996) and will consist of a sample of 350 patients who will be attended in the clinics of the Federal University of Fluminense/Institute of Health of Nova Friburgo (UFF/ISNF), in which they will be selected based on eligibility criteria. Patients aged up to 18 years, with teeth with necrotic pulps and radiographic evidence of periapical lesion will be included. These patients will be randomly divided into 8 groups: I (35 patients): unirradicular teeth will be submitted to endodontic treatment with foraminal enlargement, instrumentation with reciprocating rotation, sodium hypochlorite as irrigant, lateral condensation filling with MTA Fillapex; II (35 patients): unirradicular teeth will be submitted to endodontic treatment with foraminal enlargement, instrumentation with reciprocating rotation, sodium hypochlorite as irrigant, photobiomodulation (aPDT and LLLT), lateral condensation filling with MTA Fillapex; III (35 patients): unirradicular teeth will be submitted to endodontic treatment with foraminal enlargement, instrumentation with reciprocating rotation, chlorhexidine as irrigant, lateral condensation filling with MTA fillapex; IV (35 patients): unirradicular teeth will be submitted to endodontic treatment with foraminal enlargement, instrumentation with reciprocating rotation, sodium hypochlorite as irrigant, lateral condensation filling with AH Plus; V (35 patients): unirradicular teeth will be submitted to endodontic treatment with foraminal enlargement, instrumentation with reciprocating rotation, sodium hypochlorite as irrigant, cryotherapy with saline solution, lateral condensation filling with MTA Fillapex; VI (35 patients): unirradicular teeth will be submitted to endodontic treatment with foraminal enlargement, instrumentation with reciprocating rotation, sodium hypochlorite as irrigant, cryotherapy with saline solution, lateral condensation filling with AH Plus; VII (35 patients): unirradicular teeth will be submitted to endodontic treatment with foraminal enlargement, instrumentation with reciprocating rotation, sodium hypochlorite as irrigant, ozone therapy, lateral condensation filling with MTA Fillapex; VIII (35 patients): unirradicular teeth will be submitted to endodontic treatment with foraminal enlargement, instrumentation with reciprocating rotation, sodium hypochlorite as irrigant, ozone therapy, lateral condensation filling with AH Plus; IX (35 patients): molars will be submitted to endodontic treatment with foraminal enlargement, instrumentation with reciprocating rotation, conventional irrigation with sodium hypochlorite, lateral condensation filling with MTA fillapex; X (35 patients): molars will be submitted to endodontic treatment with foraminal enlargement, instrumentation with reciprocating rotation, passive ultrasonic irrigation with sodium hypochlorite, lateral condensation filling with MTA fillapex. The analysis of the postoperative symptoms will be performed by the visual analog pain scale at 1th, 2th, 3th, 4th, 5th, 6th, 7th, 14th and 30th days and by the clinical evaluation of edema in 48 and 72 hours. The periapical lesion repair will be evaluated clinically and radiographically at 3, 6, 12, 18 and 24 months. The longevity of rehabilitations will be performed clinically and radiographically for 24 months. In addition, patients will respond a quality of life questionnaire (OHIP-14) on the day of endodontic treatment, on the 7th day and on the 30th day.

Data analysis: The data will be inserted into a statistical program (SPSS), obtaining the frequencies of the characterization variables of the sample. The appropriate tests will be used to compare the means of the groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals over 18 years of age.
* Unirradicular teeth or molars with necrotic pulps and radiographic evidence of periapical lesion.

  * The state of the pulp will be determined by tests of sensitivity to cold and hot and confirmed by the absence of bleeding when accessing the pulp chamber.

Exclusion Criteria:

* Patients with preoperative pain.
* Patients with edema.
* Individuals with systemic disorders and pregnant.
* Positive history of antibiotic use in the last month.
* Patients who require antibiotic pre-medication for dental treatment.
* Positive history of analgesics in the previous 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2017-10-30 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain assessed by visual analog scale after endodontic treatment with enlargement of the apical foramen, in necrotic teeth and periapical lesion, and used photobiomodulation and different irrigating solutions. | Postoperative pain will be assessed by visual analog scale to measure the change of pain in first, second, third, fourth, fifth, sixth, seventh, fourteenth, and thirtieth days.
  To assess clinically the relationship of photobiomodulation and different irrigating substances (sodium hypochlorite and chlorhexidine) with or without ultrasonic activation in postoperative pain evaluated through visual analog scale, after endodontic treatment with enlargement of the apical foramen, in necrotic teeth and periapical lesion. This scale is represented by a ruler from 0 to 10, in which zero means without pain and progressively to ten, severe pain.
Edema assessed by photography after endodontic treatment with enlargement of the apical foramen, in necrotic teeth and periapical lesion, and used photobiomodulation and different irrigating solutions (sodium hypochlorite and chlorhexidine). | Edema will be evaluated by photos in 48 and 72 hours. The photo will be taken from the face to assess the edema of the region after treatment.
  To assess edema by photos after foraminal enlargement with photobiomodulation and different irrigating substances (sodium hypochlorite and chlorhexidine) with or without ultrasonic activation.

SECONDARY OUTCOMES:
Radiografic evaluation of apical repair after endodontic treatment with foraminal enlargement. | Radiographs of each tooth will be performed using a standardized digital radiograph at 3, 6, 12, 18 and 24 months. The periapical repair will be determined through radiographs as cured, in the healing process and failure.
  Carry out the radiographic follow-up of the analyzed groups for 2 years in order to show periapical healing.
Clinical and radiographic evaluation of rehabilations after endodontic treatment with foraminal enlargement. | Definitive restorations will be evaluated in adequate; inadequate and missing.
  Carry out clinical and radiographic follow-up of the groups analyzed for 2 years to demonstrate the longevity of rehabilitations. Clinical evaluation will be done through the examination of definitive restorations in adequate (any permanent restoration that appears radiographically intact); Inadequate (any permanent restoration with detectable radiographic signs of protrusions, fractured margins, recurrent caries) and missing.
Oral health-related quality of life assessed by OHIP-14, after endodontic treatment with enlargement of the apical foramen, in necrotic teeth and periapical lesion. | OHIP-14 will be performed on the day of endodontic treatment, on the 7th day and on the 30th day. This questionnaire has 14 questions in which the patient answers between never (0), rarely (1), sometimes (2), repeatedly (3) and always (4).
  To analyze the quality of life through a questionnaire (OHIP-14), before and after the endodontic treatment with foraminal enlargement in necrotic teeth and with periapical lesion. This questionnaire has 14 questions in which the patient answers between never (0), rarely (1), sometimes (2), repeatedly (3) and always (4), with maximum possible score reaching 56 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Lívia Azeredo Alves Antunes, Nova Friburgo, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided